CLINICAL TRIAL: NCT00846066
Title: Effective Educational Instruction in Preventive Oral Health: Hands On Training (HOT)Versus Web Based Training (WBT): A Randomized Control Trial
Brief Title: Oral Health Training Program for Pediatric Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Nasreen Talib, Pediatrician, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IRB# 06 10-150E
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2009-10-22 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-07

CONDITIONS: Preventive Oral Health
Keywords: educational research,; instructional methods,; Hands on training,; Web based training,; pediatric residents; preventive oral health,; dental caries,; Instructional strategies in Preventive Oral health; Web-based training on Preventive Oral Health; Hands on Training on Preventive Oral Health
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hands on Training (Experimental): Hands on Training by a pediatric dentist
  Interventions: Other: Hands on training; Other: Web based training
- Web Based Training (Active Comparator): Web Based Training for all residents before randomization
  Interventions: Other: Web based training

INTERVENTIONS:
Other: Hands on training — Hands on training by a pediatric dentist on preventive oral health
  Other Names: Active educational training with a pediatric dentist
  Arms: Hands on Training
Other: Web based training — Web based training alone
  Other Names: Educational Web Based Training for all residents

SUMMARY:
The purpose of this study was to compare the effect of the addition of hands on training by a pediatric dentist on the pediatric residents skills, confidence, opinions and practice related to preventive oral health.

DETAILED DESCRIPTION:
Objectives:

To compare the addition of Hands on Training (HOT) to Web Based Training (WBT)on residents' skills, confidence, opinions and practice .

Methods: Pediatric residents participated in WBT on preventive oral health. Then the WBT subjects were randomly assigned to receive HOT by a dentist, or WBT alone. All subjects were assessed on skills in the performance of an oral exam, by direct observation. Residents' confidence regarding oral health counseling, and their opinions about the importance of the incorporation of oral health into the well child visit, was measured by surveys utilizing a Likert scale. Residents' change in practice was assessed by a retrospective chart audit.

ELIGIBILITY:
Inclusion Criteria:

Pediatric Residents in the Continuity Care Clinics at Children's Mercy Hospital during the months of January and February 2007

Exclusion Criteria:

1. Residents on leave of absence
2. Residents who have their Continuity Care Clinics off site
3. Residents refusing consent for inclusion of results in study

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasreen J Talib, MD,MPH, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Childrens Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Pediatric residents, in the Continuity Clinic Rotation (CCC) at a general pediatric ambulatory clinic, in an urban tertiary care children's hospital, were invited to participate. Residents in any year of training were considered eligible for the study, recruitment took place in January, 2007
Pre-assignment Details: 59 participants were evaluated for the pre-test knowledge, they were next administered the Web Based Training and were then evaluated for the post-test knowledge. 56 participants were then randomized into two groups, 3 were excluded, (2 refused consent and 1 deviated from the protocol).
Groups:
- Web Based Training Only (WBT): This group received only the web based training prior to randomization(control group)
- WBT Plus Hands on Training (HOT): This group received WBT prior to randomization and additional Hands on Training by a Pediatric Dentist after randomization(intervention group)
Period: Overall Study
Arm/Group | Web Based Training Only (WBT) | WBT Plus Hands on Training (HOT)
Started | 27 | 29
Completed | 27 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- WBT Only: Control Group Web Based Training only
- WBT+HOT: Web Based Training plus Hands on Training
- Total: Total of all reporting groups
Arm/Group | WBT Only | WBT+HOT | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 29 | 56
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 8 | 6 | 14
Level of Training [Number; unit: participants] — The level of training during residency,
  participants
    First year Residents | 12 | 11 | 23
    Second and Third year Residents | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Correct Skills
Description: Skills were observed by pediatric dentists for each resident utilizing a six item checklist 3 months after the intervention (HOT) was completed.Each correct skill demonstrated was scored as 1 (16.67%) with a maximum of 6 representing 100%.The mean pecentage of correct skills were measured by direct observation by a pediatric dentist among the WBT alone and WBT+HOT groups
Time Frame: 3 months after Hands-on Training (HOT)
Measure: Mean (Standard Deviation); unit: Percentage of correct skills
Arm/Group | WBT Only | WBT+HOT
Number analyzed (Participants) | 27 | 29
Percentage of correct skills | 73 (27) | 87 (21)

2. Primary Outcome: Percent Change From Baseline in Confidence at 4 Months
Description: Confidence was measured by self-administered surveys regarding knowledge and practice of oral health. The surveys used a 4 point Likert scale (1=not confident, 4=very confident).The mean percent of change in the responses of "very confident" was compared between both groups. The percentage change equals {(mean score at 4 months-mean score at baseline)/ mean score at baseline} *100%
Time Frame: Baseline and 4 months
Population: Only completed paired (pre/post intervention) surveys were analyzed
Measure: Mean (Standard Deviation); unit: Percent change.
Groups:
- WBT + HOT: Web Based Training plus Hands on Training
Arm/Group | WBT Only | WBT + HOT
Number analyzed (Participants) | 22 | 19
Percent change. | 14 (.33) | 19 (.38)

3. Primary Outcome: Percent Change From Baseline in Opinions Regarding Incorporating Oral Health Into a Well Child Visit at 4 Months
Description: Opinions regarding incorporating oral health into a well child visit was measured by self administered surveys. The surveys used a 4 point Likert scale from 1 for (strongly disagree) to 4 for (strongly agree). Mean percentage change in the "agree" and "strongly agree" responses by the residents was compared between both groups. The percentage change equals {(mean score at 4 months-mean score at baseline)/ mean score at baseline} *100%
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | WBT Only | WBT+HOT
Number analyzed (Participants) | 27 | 29
Percent change | -11 (.33) | -33 (.42)

4. Primary Outcome: Percent Change From Baseline in Practice of Oral Health Based on Pre and Post Study Chart Audit at 6 Months
Description: The mean percent change in the documentation of oral health components at a well child visit. This was done by an audit of a random selection of 5 charts of patients who came in for well child visits, completed by each resident at baseline and at 6 months later.We scored this utilizing a 4 item checklist each correct item was scored as 1 (25%), with a maximum of 4(100%). The percentage change used the following formula {(mean score at 6 months-mean score at baseline)/mean score at baseline}*100%
Time Frame: At baseline and 6 months
Population: Analysis per protocol. Subjects dropped from analysis because charts not available within the time frame of the study and incomplete data.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | WBT Only | WBT+HOT
Number analyzed (Participants) | 19 | 18
Percent change | 26.32 (13.25) | 36.67 (22.42)

ADVERSE EVENTS:
Description: Total number of Participants Risk is 0. This is because serious and other non serious adverse events were not collected or assessed. This was an educational intervention
Arm/Group | Web Based Training Only (WBT) | WBT Plus Hands on Training (HOT)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes